CLINICAL TRIAL: NCT06962046
Title: Can the Use of Virtual Reality Improve Outcomes Following Total Knee Arthroplasty With Spinal Anaesthesia? - A Pilot Study
Brief Title: Can the Use of Virtual Reality Improve TKA Outcomes
Acronym: VR-TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19066DJ-SW
Record Dates: First submitted 2024-08-28; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-01

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: A single centred, parallel group, randomised controlled tria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality (Experimental)
  Interventions: Procedure: Virtual Reality
- Control (No Intervention): Standard Care

INTERVENTIONS:
Procedure: Virtual Reality — * VR
  * Spinal anaesthesia
  * Limited propofol aiming for OAA/S of 4-5 (light sedation)
  Arms: Virtual Reality

SUMMARY:
Virtual reality (VR) uses computer technology to create a three-dimensional environment which the user can explore and interact with. VR can be used to distract the patient during an operation and has been used to avoid sedative premedication, increase patient satisfaction and decrease pain during nerve blocks. VR used alongside spinal anaesthetic for hip, knee and ankle operations has shown a trend of less sedation being required with no decrease in patient satisfaction.

The most common type of anaesthesia given during total knee arthroplasty (TKA) is spinal. Spinal anaesthesia is given unless there are complications or other conditions present, and general anaesthesia is given instead. General anaesthesia puts the patient to sleep during the operation, whereas spinal anaesthesia allows the patient to stay awake, but numbs the lower half of the body so no pain is felt. Sedation is usually given with spinal anaesthesia to make the patient relaxed and sleepy. Light sedation will allow the patient to be awake but relaxed, whereas deeper sedation means the patient is more likely to be asleep and less likely to recall what happened during the operation. Sedation can cause a number of side effects including nausea, vomiting, headache, drowsiness, pain, confusion, memory loss and breathing difficulties.

In this study, all patients will receive spinal anaesthesia. Group 1 will receive VR and a light level of sedation, whilst Group 2 will not receive VR but will receive a deeper level of sedation (standard of care). When using VR during TKA, a lighter level of sedation should be required. This could help to reduce side effects and aid quicker patient recovery. This pilot study aims to investigate this further.

DETAILED DESCRIPTION:
Total joint arthroplasty (TJA) is a successful surgical intervention to reduce pain and immobility from osteoarthritis. Mortality rates following TJA are low and survival has been increasing over the last two and a half decades despite an ageing population with a higher frequency of comorbidities.

Perioperative virtual reality (VR) is a non-pharmacological technique which has been used effectively to avoid sedative pre-medication, increase patient satisfaction and alleviate procedural pain during nerve blocks. VR has been successfully utilised across different medical specialties to reduce patient anxiety associated with interventions including magnetic resonance imaging (MRI), physical therapy, dental pain, and change of burns dressings. Furthermore, a trend towards less propofol sedation with use of VR has been found in spinal anaesthetic for hip, knee and ankle operations, with no decrease in patient satisfaction. However, this small pilot study did not investigate any other outcomes other than type and amount of sedation and duration of surgery. VR use has also been shown to reduce fentanyl dose, midazolam use and pain in elective total knee arthroplasty (TKA) patients who received a pre-operative adductor canal catheter. Satisfaction of patient, surgeon and anaesthetist has also been compared when using VR and using sedation with midazolam in patients undergoing urologic surgery under spinal anaesthesia. The patient and anaesthetist satisfaction scores were significantly higher in the VR group than in the sedation group.

Sedation is associated with a number of post-operative complications including nausea, hypo/hypertension, lower respiratory tract infection, cardiac arrhythmias, peripheral nerve damage, and post-operative delirium (PD). Nausea is a common occurrence following surgery with reported incidences of 30% in all post-surgical patients and up to 80% in high-risk patients. Dose dependent hypotension is the common complication in patients who have received propofol sedation, particularly in volume depleted patients. A common cardiovascular complication during anaesthesia is arrhythmia, with 70% of patients having arrhythmia undergoing general anaesthesia for various surgical procedures. Further complications associated with propofol, although more uncommon, include hypertriglyceridemia, pancreatitis and allergic complications.

The incidence of PD is generally higher after hip fracture surgery (4-53.3%) compared to elective hip surgery (3.6-28.3%). Independent risk factors for developing inpatient delirium include dementia, age, visual impairment, functional impairment and increased comorbidities. While most studies measuring effect of propofol on sleep disturbance and PD have focussed on the critical care setting, light propofol sedation (to target a bispectral index (BIS) >80) decreased the prevalence of PD by 50% compared to deep sedation (BIS target of 50) in patients undergoing hip surgery with spinal anaesthesia. A further RCT investigated whether limiting propofol sedation with spinal anaesthesia in non-elective hip fracture repair patients reduced risk of delirium post-operatively. Patients were randomised to receive either heavier sedation (modified observer's assessment of alertness/sedation score (OAA/S) of 0-2) or lighter sedation (OAA/S of 4-5). There were no significant differences in risk of incident delirium between the heavier and lighter sedation groups. However, when stratified by Charlson comorbidity index (CCI), in low comorbid states, heavier sedation levels doubled the risk of delirium compared to lighter sedation. This randomised controlled trial (RCT) recruited hip fracture patients with a mean age of 82 years. Therefore, a similar study should be conducted in younger, less comorbid patients undergoing elective joint arthroplasty.

Sedation can also affect recovery following surgery. Being male, nausea, vomiting and pain during the ward stay have been reported to be risk factors for poor quality of recovery after sedation with midazolam for lower limb orthopaedic surgeries. Poor quality of recovery following surgery can also increase hospital stay and health care resources. No significant difference in quality of recovery has been reported between those who experienced immersive VR and those who underwent conventional care.

Propofol infusions are commonly administered alongside spinal anaesthesia for orthopaedic surgery. It is commonly given with no specific objective clinical target end point. This gives rise to the potential of administering excess propofol which may result in inadvertent deep levels of sedation. This can cause prolonged periods of inadvertent general anaesthesia depth during 'regional' cases (often without insertion of an airway device). Therefore, it is important to investigate potential ways of lowering propofol infusions during surgery, without increasing patient risk, anxiety or pain, such as through the use of VR.

Aims of Study

The aims of this pilot study are to determine:

1. the feasibility of using VR during TKA with spinal anaesthesia.
2. what outcomes, if any, can be influenced using VR during TKA with spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old who are American Society of Anaesthesiologists (ASA) grade 1 or 2 scheduled for routine primary elective knee arthroplasty.

Exclusion Criteria:

* Patients who are ASA grade 3 or 4.
* Patients who cannot use VR e.g. those with dementia.
* Patients with an existing diagnosis of delirium.
* Patients with visual impairment if degree of myopia/hyperopia exceeds the corrective power of the VR headset.
* Patients with hearing aids.
* Patients with previous history of motion sickness.
* Patients with epilepsy, history of black outs or fitting.
* Patients who will have an operation over 1 hour in duration or any patient who requires more complex surgery.
* Patients who have requested no sedation during the operation.
* Patients who have received premedication.
* Patients who have a general anaesthetic.
* Patients who do not adequately understand verbal explanations or written information given in English, or who have special communication needs.
* Patients who are not capable of informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using VR during total knee arthroplasty with spinal anaesthesia | Postoperative Day 1
  Feasibility of using VR during total knee arthroplasty will be assessed by recruitment numbers to the study and staff and patients will be asked for their views of using the VR equipment.

SECONDARY OUTCOMES:
4AT | 1 hour, 24 hours and 48 hours following skin closure.
  The 4AT includes alertness, Abbreviated Mental Test 4 (AMT4), attention and acute change or fluctuating course. A score of 4 or above indicates possible delirium and/or cognitive impairment, a score of 1-3 indicates possible cognitive impairment and a score of 0 indicates that delirium or severe cognitive impairment is unlikely.
Logical Memory subtest of the WMS-IV UK | 1 hour and 24 hours following skin closure.
  The Logical Memory subtest of the WMS-IV UK will be used to assess memory recall pre-operatively, at 1 hour (+/- 30 minutes) in recovery and at 24 hours (+/- 2 hours) following skin closure. Logical Memory I assesses narrative memory under a free recall condition. Logical Memory II is a delayed condition assessing long-term narrative memory with free recall and recognition tasks.
Total Propofol during operation | 1 hour following skin closure.
  Total propofol administered during the operation will be recorded in mg/kg.
E-entropy | 1 hour following skin closure.
  The e-entropy system uses a disposable 4-electrode sensor on the patient&amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;#39;s forehead to measure electrical activity in the brain before using a proprietary algorithm to process the electroencephalogram data and calculate a number between 0 (absence of brain electrical activity) and 100 (wide awake) providing an objective measure of the patient's depth of consciousness. The average e-entropy score during the operation will be recorded by calculating a mean of the trend data from the monitor log.
Discharge from Recovery | Every 15 minutes in recovery up until 2 hours.
  The time until ready for discharge from recovery will be recorded using the NEWS criteria. The time point that the following objectives are met will also be recorded; spinal regression below T4, temperature ≥36 degrees, pain score &amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;lt;3, nausea score between 0-1 and NEWS criteria ≤ 3.
Mobilisation | 4 hours following skin closure.
  Mobilisation will be assessed by a physiotherapist using the Timed Up and Go (TUG) test at 4 hours (+/- 1 hour) following skin closure. This will be recorded as the time in seconds which it takes a patient to stand up from a chair with armrests, walk 3 metres at a comfortable and safe pace, turn, walk back to the chair and sit back down again.
Quality of Recovery | 4 hours (+/- 1 hour) and at 24 hours (+/- 2 hours) following skin closure.
  Quality of recovery will be measured using the Quality of Recovery (QoR)-15 survey (Appendix 4) at 4 hours (+/- 1 hour) and at 24 hours (+/- 2 hours) following skin closure. The QoR-15 score ranges from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery).
IV fluids | Up to 1 week post operation.
  Total IV fluids will be measured in ml/kg for the duration of the patient's hospital stay.
Length of stay | Up to 1 week post operation.
  Total length of stay will be calculated using date of discharge and date of operation.
Post-operative analgesia | Up to 1 week post operation.
  Patient notes will be assessed retrospectively for post-operative analgesia. Type and total dose of analgesia taken on each post operative 24 hour period up until discharge or up until 1 week post operation will be recorded.
Anti-emetic use | Up to 1 week post operation.
  Patient notes will be assessed retrospectively for anti-emetic use. Type and total dose of anti-emetics taken on each post operative 24 hour period up until discharge or up until 1 week post operation will be recorded.
Any inpatient complications | Up to 1 week post operation.
  Patient notes will be assessed retrospectively for any inpatient complications including vasovagal, fall, arrthymia, bleed, take back, and escalation of care.

CONTACTS AND LOCATIONS:
Overall Officials: David Johnston, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Musgrave Park Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamel MB, Toth M, Legedza A, Rosen MP. Joint replacement surgery in elderly patients with severe osteoarthritis of the hip or knee: decision making, postoperative recovery, and clinical outcomes. Arch Intern Med. 2008 Jul 14;168(13):1430-40. doi: 10.1001/archinte.168.13.1430. PMID 18625924
- [Background] Lalmohamed A, Vestergaard P, de Boer A, Leufkens HG, van Staa TP, de Vries F. Changes in mortality patterns following total hip or knee arthroplasty over the past two decades: a nationwide cohort study. Arthritis Rheumatol. 2014 Feb;66(2):311-8. doi: 10.1002/art.38232. PMID 24504803
- [Background] Bekelis K, Calnan D, Simmons N, MacKenzie TA, Kakoulides G. Effect of an Immersive Preoperative Virtual Reality Experience on Patient Reported Outcomes: A Randomized Controlled Trial. Ann Surg. 2017 Jun;265(6):1068-1073. doi: 10.1097/SLA.0000000000002094. PMID 27906757
- [Background] Pandya PG, Kim TE, Howard SK, Stary E, Leng JC, Hunter OO, Mariano ER. Virtual reality distraction decreases routine intravenous sedation and procedure-related pain during preoperative adductor canal catheter insertion: a retrospective study. Korean J Anesthesiol. 2017 Aug;70(4):439-445. doi: 10.4097/kjae.2017.70.4.439. Epub 2017 Mar 15. PMID 28794840
- [Background] Brown RKJ, Petty S, O'Malley S, Stojanovska J, Davenport MS, Kazerooni EA, Fessahazion D. Virtual Reality Tool Simulates MRI Experience. Tomography. 2018 Sep;4(3):95-98. doi: 10.18383/j.tom.2018.00023. PMID 30320208
- [Background] Ashmore J, Di Pietro J, Williams K, Stokes E, Symons A, Smith M, Clegg L, McGrath C. A Free Virtual Reality Experience to Prepare Pediatric Patients for Magnetic Resonance Imaging: Cross-Sectional Questionnaire Study. JMIR Pediatr Parent. 2019 Apr 18;2(1):e11684. doi: 10.2196/11684. PMID 31518319
- [Background] Carrougher GJ, Hoffman HG, Nakamura D, Lezotte D, Soltani M, Leahy L, Engrav LH, Patterson DR. The effect of virtual reality on pain and range of motion in adults with burn injuries. J Burn Care Res. 2009 Sep-Oct;30(5):785-91. doi: 10.1097/BCR.0b013e3181b485d3. PMID 19692911
- [Background] Furman E, Jasinevicius TR, Bissada NF, Victoroff KZ, Skillicorn R, Buchner M. Virtual reality distraction for pain control during periodontal scaling and root planing procedures. J Am Dent Assoc. 2009 Dec;140(12):1508-16. doi: 10.14219/jada.archive.2009.0102. PMID 19955069
- [Background] Mott J, Bucolo S, Cuttle L, Mill J, Hilder M, Miller K, Kimble RM. The efficacy of an augmented virtual reality system to alleviate pain in children undergoing burns dressing changes: a randomised controlled trial. Burns. 2008 Sep;34(6):803-8. doi: 10.1016/j.burns.2007.10.010. Epub 2008 Mar 5. PMID 18325675
- [Background] Chan PY, Scharf S. Virtual Reality as an Adjunctive Nonpharmacological Sedative During Orthopedic Surgery Under Regional Anesthesia: A Pilot and Feasibility Study. Anesth Analg. 2017 Oct;125(4):1200-1202. doi: 10.1213/ANE.0000000000002169. PMID 28598921
- [Background] Moon JY, Shin J, Chung J, Ji SH, Ro S, Kim WH. Virtual Reality Distraction during Endoscopic Urologic Surgery under Spinal Anesthesia: A Randomized Controlled Trial. J Clin Med. 2018 Dec 20;8(1):2. doi: 10.3390/jcm8010002. PMID 30577461
- [Background] Inverso G, Dodson TB, Gonzalez ML, Chuang SK. Complications of Moderate Sedation Versus Deep Sedation/General Anesthesia for Adolescent Patients Undergoing Third Molar Extraction. J Oral Maxillofac Surg. 2016 Mar;74(3):474-9. doi: 10.1016/j.joms.2015.10.009. Epub 2015 Oct 16. PMID 26546845
- [Background] Amornyotin S. Sedation-related complications in gastrointestinal endoscopy. World J Gastrointest Endosc. 2013 Nov 16;5(11):527-33. doi: 10.4253/wjge.v5.i11.527. PMID 24255744
- [Background] De Gaudio AR, Rinaldi S. Sedation in PACU: indications, monitoring, complications. Curr Drug Targets. 2005 Nov;6(7):729-40. doi: 10.2174/138945005774574542. PMID 16305450
- [Background] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557
- [Background] Sieber FE, Neufeld KJ, Gottschalk A, Bigelow GE, Oh ES, Rosenberg PB, Mears SC, Stewart KJ, Ouanes JP, Jaberi M, Hasenboehler EA, Li T, Wang NY. Effect of Depth of Sedation in Older Patients Undergoing Hip Fracture Repair on Postoperative Delirium: The STRIDE Randomized Clinical Trial. JAMA Surg. 2018 Nov 1;153(11):987-995. doi: 10.1001/jamasurg.2018.2602. PMID 30090923
- [Background] Marik PE. Propofol: therapeutic indications and side-effects. Curr Pharm Des. 2004;10(29):3639-49. doi: 10.2174/1381612043382846. PMID 15579060
- [Background] Kwon CH, Kim SH. Intraoperative management of critical arrhythmia. Korean J Anesthesiol. 2017 Apr;70(2):120-126. doi: 10.4097/kjae.2017.70.2.120. Epub 2017 Feb 21. PMID 28367281
- [Background] Sharma PT, Sieber FE, Zakriya KJ, Pauldine RW, Gerold KB, Hang J, Smith TH. Recovery room delirium predicts postoperative delirium after hip-fracture repair. Anesth Analg. 2005 Oct;101(4):1215-1220. doi: 10.1213/01.ane.0000167383.44984.e5. PMID 16192548
- [Background] Bitsch MS, Foss NB, Kristensen BB, Kehlet H. Acute cognitive dysfunction after hip fracture: frequency and risk factors in an optimized, multimodal, rehabilitation program. Acta Anaesthesiol Scand. 2006 Apr;50(4):428-36. doi: 10.1111/j.1399-6576.2005.00899.x. PMID 16548854
- [Background] Bruce AJ, Ritchie CW, Blizard R, Lai R, Raven P. The incidence of delirium associated with orthopedic surgery: a meta-analytic review. Int Psychogeriatr. 2007 Apr;19(2):197-214. doi: 10.1017/S104161020600425X. Epub 2006 Sep 14. PMID 16973101
- [Background] Inouye SK, Zhang Y, Jones RN, Kiely DK, Yang F, Marcantonio ER. Risk factors for delirium at discharge: development and validation of a predictive model. Arch Intern Med. 2007 Jul 9;167(13):1406-13. doi: 10.1001/archinte.167.13.1406. PMID 17620535
- [Background] Moro ET, Silva MA, Couri MG, Issa DD, Barbieri JM. Quality of recovery from anesthesia in patients undergoing orthopedic surgery of the lower limbs. Braz J Anesthesiol. 2016 Nov-Dec;66(6):642-650. doi: 10.1016/j.bjane.2015.05.001. Epub 2016 Sep 30. PMID 27793240
- [Background] Liu J, Yuan W, Wang X, Royse CF, Gong M, Zhao Y, Zhang H. Peripheral nerve blocks versus general anesthesia for total knee replacement in elderly patients on the postoperative quality of recovery. Clin Interv Aging. 2014 Feb 18;9:341-50. doi: 10.2147/CIA.S56116. eCollection 2014. PMID 24600214
- [Background] Sieber FE, Gottshalk A, Zakriya KJ, Mears SC, Lee H. General anesthesia occurs frequently in elderly patients during propofol-based sedation and spinal anesthesia. J Clin Anesth. 2010 May;22(3):179-83. doi: 10.1016/j.jclinane.2009.06.005. PMID 20400003
- [Background] Bellelli G, Morandi A, Davis DH, Mazzola P, Turco R, Gentile S, Ryan T, Cash H, Guerini F, Torpilliesi T, Del Santo F, Trabucchi M, Annoni G, MacLullich AM. Validation of the 4AT, a new instrument for rapid delirium screening: a study in 234 hospitalised older people. Age Ageing. 2014 Jul;43(4):496-502. doi: 10.1093/ageing/afu021. Epub 2014 Mar 2. PMID 24590568
- [Background] Singh H. Bispectral index (BIS) monitoring during propofol-induced sedation and anaesthesia. Eur J Anaesthesiol. 1999 Jan;16(1):31-6. doi: 10.1046/j.1365-2346.1999.00420.x. PMID 10084098
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Myles PS, Reeves MD, Anderson H, Weeks AM. Measurement of quality of recovery in 5672 patients after anaesthesia and surgery. Anaesth Intensive Care. 2000 Jun;28(3):276-80. doi: 10.1177/0310057X0002800304. PMID 10853209
- See also: National Early Warning Score (NEWS) — https://www.mdcalc.com/calc/1873/national-early-warning-score-news
- See also: Pearson Education Ltd. Wechsler Memory Scale - Fourth UK Edition (WMS-IV UK). — https://www.pearsonclinical.co.uk/store/ukassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Wechsler-Memory-Scale---Fourth-UK-Edition/p/P100009265.html